CLINICAL TRIAL: NCT00422383
Title: A Randomized, Double-blind Study to Evaluate the Effect of Various Re-treatment Regimens of MabThera in Combination With Methotrexate on Treatment Response in Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate.
Brief Title: A Study of Retreatment With MabThera (Rituximab) in Combination With Methotrexate in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA17044
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]
- 2 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]
- 3 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 500mg iv in days 1 and 15, and 500mg iv on days 168 and 182
  Arms: 1
Drug: rituximab [MabThera/Rituxan] — 500mg iv on days 1 and 15, and 1000mg iv on days 168 and 182
  Arms: 2
Drug: rituximab [MabThera/Rituxan] — 1000mg iv on days 1 and 15 and 1000mg iv (or placebo in UK)on days 168 and 182
  Arms: 3

SUMMARY:
This study will evaluate the efficacy and safety of various treatment and retreatment regimens of MabThera. All patients will receive concomitant methotrexate, 10-25mg once weekly either orally or parenterally. The anticipated time on study treatment is 2+ years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* RA for >=6 months;
* receiving outpatient treatment;
* inadequate response to methotrexate, having received and tolerated it for >=12 weeks, with a stable dose for >=4 weeks.

Exclusion Criteria:

* rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA;
* inflammatory joint disease other than RA, or other systemic autoimmune disorder;
* diagnosis of juvenile arthritis, or RA before the age of 16;
* previous treatment with >1 biologic agent, any cell-depleting therapies, or concurrent treatment with any biologic agent or DMARD other than methotrexate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2006-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (85):
- Australia (6):
  - Coffs Harbour, New South Wales
  - Sydney, New South Wales
  - Maroochydore, Queensland
  - Southport, Queensland
  - Malvern, Victoria
  - Melbourne, Victoria
- Ghent, Belgium
- Brazil (2):
  - Goiânia, Goiás
  - São Paulo, São Paulo
- Canada (7):
  - Penticton, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Trois-Rivières, Quebec
- Beijing, China
- Oulu, Finland
- France (8):
  - Bois-Guillaume
  - Bordeaux
  - Dijon
  - Le Mans
  - Lille
  - Montpellier
  - Nice
  - Paris
- Germany (7):
  - Bad Nauheim
  - Cologne
  - Hamburg
  - Heidelberg
  - Herne
  - Osnabrück
  - Ratingen
- Hungary (2):
  - Debrecen
  - Eger
- Italy (13):
  - Coppito, Abruzzo
  - Potenza, Basilicate
  - Ferrara, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Arenzano, Liguria
  - Genoa, Liguria
  - Pieve di Coriano, Lombardy
  - Turin, Piedmont
  - Palermo, Sicily
  - Pisa, Tuscany
  - Prato, Tuscany
  - Siena, Tuscany
  - Valeggio sul Mincio, Veneto
- Netherlands (3):
  - Amsterdam
  - Leiden
  - Nijmegen
- New Zealand (3):
  - Auckland
  - Christchurch
  - Timaru
- Slovakia (2):
  - Košice
  - Piešťany
- South Africa (3):
  - Cape Town
  - Diepkloof
  - Pretoria
- Spain (6):
  - Barcelona, Barcelona
  - Burgos, Burgos
  - León, Leon
  - Madrid, Madrid
  - Gijón, Principality of Asturias
  - Seville, Sevilla
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- United Kingdom (14):
  - Barnsley
  - Birmingham
  - Cambridge
  - Glasgow
  - London
  - Londonderry
  - Manchester
  - Metropolitan Borough of Wirral
  - Middlesbrough
  - Northampton
  - Nottingham
  - Reading
  - Truro
  - Wigan

REFERENCES:
- [Derived] Rubbert-Roth A, Tak PP, Zerbini C, Tremblay JL, Carreno L, Armstrong G, Collinson N, Shaw TM; MIRROR Trial Investigators. Efficacy and safety of various repeat treatment dosing regimens of rituximab in patients with active rheumatoid arthritis: results of a Phase III randomized study (MIRROR). Rheumatology (Oxford). 2010 Sep;49(9):1683-93. doi: 10.1093/rheumatology/keq116. Epub 2010 May 12. PMID 20463186

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Low Dose Plus (+) Methotrexate: Participants received rituximab, 0.5 grams (g), intravenously (IV), on Days 1, 15, 168, and 182. Participants also received methylprednisolone 100 milligrams (mg), IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 milligrams per milliliter (mg/mL), orally (PO) or parenterally, as prescribed. Participants also received a stable dose of folate greater than or equal to (≥) 5 milligrams per week (mg/week) given either as a single dose or as a divided weekly dose.
- Rituximab Escalated Dose + Methotrexate: Participants received rituximab, 0.5 g, IV, on Days 1 and 15 and 1.0 g, IV, on Days 168 and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parenterally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose.
- Rituximab High Dose + Methotrexate: Participants received rituximab, 1.0 g, IV, on Days 1, 15, 168, and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parenterally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose.
- Rituximab/Placebo + Methotrexate: Participants received rituximab, 1.0 g, IV, on Days 1 and 15, and a placebo, IV, on Days 168 and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parenterally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose. This treatment group was not part of the planned analysis and was not analyzed for all outcomes measures since they did not receive the planned treatment.
- Rituximab Decreased Dose + Methotrexate: Participants received rituximab, 1.0 g, IV, on Days 1 and 15 and 0.5 g, IV, on Days 168 and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parenterally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose. This treatment group was not part of the planned analysis and was not analyzed for all outcomes measures since they did not receive the planned treatment.
Period: Overall Study
Arm/Group | Rituximab Low Dose Plus (+) Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Started | 134 | 120 | 93 | 6 | 25
Completed | 119 | 106 | 89 | 4 | 22
Not Completed | 15 | 14 | 4 | 2 | 3
Not completed — Adverse Event | 5 | 3 | 1 | 1 | 0
Not completed — Lack of Efficacy | 4 | 4 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat-modified 2 (ITT-M2) population included all randomized participants who received at least 1 infusion of study treatment. Due to a UK protocol amendment error, 6 participants incorrectly received placebo. Due to medication list error, 25 participants received an incorrect dose of treatment. Participants were analyzed as treated.
Groups:
- Rituximab Low Dose + Methotrexate: Participants received rituximab, 0.5 g, IV, on Days 1, 15, 168, and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parenterally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose.
- Total: Total of all reporting groups
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate | Total
Number analyzed (Participants) | 134 | 119 | 93 | 6 | 25 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.58 (12.805) | 52.32 (12.115) | 51.26 (12.179) | 51.83 (6.274) | 52.32 (8.882) | 52.48 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 90 | 77 | 4 | 16 | 297
  Male | 24 | 29 | 16 | 2 | 9 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response as Determined by American College of Rheumatology (ACR) 20% Improvement (ACR20)
Description: ACR20 defined as overall score of ≥20 in ACR number (ACRn) calculation. Overall score defined as lowest percent improvement from baseline (BL) of following 3 measures: tender joint count (TJC; 68 joints), swollen joint count (SJC: 66 joints), and the 3rd lowest improvement achieved by at least 3 of 5 remaining ACR core parameters: physician's global assessment of disease activity, participant's global assessment of disease activity, participant's assessment of pain (visual analog assessment [VAS]), Health Assessment Questionnaire (HAQ), and C-Reactive Protein (CRP). If CRP missing, erythrocyte sedimentation rate (ESR) was used. In order for improvements in the ACRn score to be expressed as a positive result, rather than the negative changes that improvements represent, the final ACRn results were multiplied by negative 1. Last observation carried forward (LOCF) for TJC/SJC, HAQ, CRP/ESR, VAS. If change in CRP incalculable, change in ESR used. ACR20 set to Non-Responder if ACRn missing
Time Frame: Week 48
Population: ITT-M2 population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 134 | 119 | 93
percentage of participants | 64.2 [56.0 to 72.0] | 63.9 [55.0 to 72.0] | 72.0 [63.0 to 81.0]
Statistical Analysis 1: Comparison: Rituximab Low Dose + Methotrexate vs Rituximab Escalated Dose + Methotrexate; Test type: Superiority or Other; p = 0.8156, Cochran-Mantel-Haenszel; Weighted Difference = -0.01, 95% CI 2-sided [-0.13 to 0.10] — Analysis stratified by region, prior biologic use, rheumatoid factor (RF) status, and treatment
Statistical Analysis 2: Comparison: Rituximab Low Dose + Methotrexate vs Rituximab High Dose + Methotrexate; Test type: Superiority or Other; p = 0.2419, Cochran-Mantel-Haenszel; Weighted Difference = 0.07, 95% CI 2-sided [-0.05 to 0.19] — Analysis stratified by region, prior biologic use, RF status, and treatment

2. Secondary Outcome: Percentage of Participants With ACR 50% Improvement Criteria (ACR50) Response at Week 48
Description: ACR50 was defined as an overall score of 50 in the ACRn calculation. Overall score defined as lowest percent improvement from BL of following 3 measures: TJC (68 joints), SJC (66 joints), and the 3rd lowest improvement achieved by at least 3 of 5 remaining ACR core parameters: physician's global assessment of disease activity, participant's global assessment of disease activity, participant's assessment of pain (VAS), HAQ, and CRP. If CRP missing, ESR was used. In order for improvements in the ACRn score to be expressed as a positive result, rather than the negative changes that improvements represent, the final ACRn results were multiplied by negative 1. LOCF for TJC/SJC, HAQ, CRP/ESR, VAS. If change in CRP incalculable, change in ESR used. ACR50 set to Non-Responder if ACRn missing.
Time Frame: Week 48
Population: ITT-M2 population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 134 | 119 | 93
percentage of participants | 39 | 39 | 48

3. Secondary Outcome: Percentage of Participants With a ACR 70% Improvement Criteria (ACR70) Response at Week 48
Description: ACR70 was defined as an overall score of 70 in the ACRn calculation. The Overall score defined as lowest percent improvement from BL of following 3 measures: TJC (68 joints), SJC (66 joints), and the 3rd lowest improvement achieved by at least 3 of 5 remaining ACR core parameters: physician's global assessment of disease activity, participant's global assessment of disease activity, participant's assessment of pain (VAS), HAQ, and CRP. If CRP missing, ESR was used. In order for improvements in the ACRn score to be expressed as a positive result, rather than the negative changes that improvements represent, the final ACRn results were multiplied by negative 1. LOCF for TJC/SJC, HAQ, CRP/ESR, VAS. If change in CRP incalculable, change in ESR used. ACR70 set to Non-Responder if ACRn missing.
Time Frame: Week 48
Population: ITT-M2 population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 134 | 119 | 93
percentage of participants | 20 | 19 | 23

4. Secondary Outcome: Disease Activity Score Based on 28-Joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR): Adjusted Mean Change From BL at Week 48
Description: DAS28 was calculated according to the following formula: DAS28 equals (=) [0.56 multiplied by (*) the square root (√) of TJC] plus (+) [0.28 * √ of SJC] + (0.70 * the natural logarithm (ln) ESR in millimeters per hour (mm/h)] + [0.014 * participant's global assessment of disease activity (GH)]. DAS28-ESR ≥ 5.1 = high disease activity, DAS28-ESR less than or equal to (≤) 3.2 = low disease activity, DAS28-ESR less than (<) 2.6 = remission.
Time Frame: BL, Week 48
Population: ITT-M2 population. Two participants from the Low Dose group and 1 participant from the Escalated Dose group were not evaluated for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 132 | 118 | 93
score on a scale | -2.13 [-2.38 to -1.87] | -2.19 [-2.45 to -1.92] | -2.42 [-2.71 to -2.12]
Statistical Analysis 1: Comparison: Rituximab Low Dose + Methotrexate vs Rituximab Escalated Dose + Methotrexate; Test type: Superiority or Other; p = 0.7127, ANOVA — Stratified by region, prior biologic use, RF status and treatment
Statistical Analysis 2: Comparison: Rituximab Low Dose + Methotrexate vs Rituximab High Dose + Methotrexate; Test type: Superiority or Other; p = 0.1018, ANOVA — Stratified by region, prior biologic use, RF status and treatment

5. Secondary Outcome: Percentage of Participants With a Response at Week 48 by European League Against Rheumatism (EULAR) Category
Description: EULAR responses were categorized according to DAS28-ESR score. DAS28-ESR ≤ 3.2 at Week 48 and a change from BL to Week 48 < -1.2 = good response, DAS28-ESR ≤ 3.2 or greater than (>) 3.2 and ≤ 5.1 at Week 48 and a change from BL to Week 48 < -0.6 and ≥ -1.2 = moderate response, DAS28-ESR > 3.2 and ≤ 5.1 at Week 48 and a change from BL to Week 48 < -1.2 = moderate response, DAS28-ESR > 5.1 at Week 48 and a change from BL to Week 48 < -1.2 = moderate response, DAS28-ESR ≤ 3.2 or > 3.2 and ≤ 5.1 at Week 48 and a change from BL to Week 48 ≥ -0.6 = no response, DAS28-ESR > 5.1 at Week 48 and a change from BL to Week 48 < -0.6 and ≥ -1.2 or ≥ -0.6 = no response.
Time Frame: Week 48
Population: ITT-M2 population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 134 | 119 | 93
percentage of participants
  None | 26.9 | 27.7 | 10.8
  Moderate | 50.7 | 55.5 | 62.4
  Good | 22.4 | 16.8 | 26.9
Statistical Analysis 1: Comparison: Rituximab Low Dose + Methotrexate vs Rituximab Escalated Dose + Methotrexate; Test type: Superiority or Other; p = 0.5029, Cochran-Mantel-Haenszel — Stratified by region, prior biologic use, RF status, and treatment
Statistical Analysis 2: Comparison: Rituximab Low Dose + Methotrexate vs Rituximab High Dose + Methotrexate; Test type: Superiority or Other; p = 0.0495, Cochran-Mantel-Haenszel — Stratified by region, prior biologic use, RF status, and treatment

6. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score From BL at Week 48
Description: FACIT-F scores were obtained from a 13 question self-administered participant questionnaire designed to measure the degree of fatigue experienced by participants in the previous 7 days. Participants responded to the questions using a value between 0 and 4, where 0 indicated "not at all" and 4 indicated "very much." 11 of the 13 questions were negatively stated; indicating the higher the score of the participant's response, the greater their fatigue. These questions were calculated as 4 minus the participants' response, so that a higher score indicated an improvement in health. The scores for the 2 positively stated questions were not changed. The participants' responses were summed to result in an overall score, which are scored 0 to 52 (52 = highest level of functioning). A positive change from BL indicated improvement.
Time Frame: BL, Week 48
Population: ITT-M2 population. 9, 4, 2, and 1 participants were not evaluated for this outcome measure from the Low Dose, Escalated Dose, High Dose, and Decreased Dose groups, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 125 | 115 | 91 | 6 | 24
score on a scale | 6.605 (10.1529) | 8.109 (10.2876) | 8.364 (9.8368) | 2.000 (16.0250) | 6.192 (12.0081)

7. Secondary Outcome: Short-Form 36 Health Survey (SF-36) Score
Description: SF-36 scores were obtained by scoring participants' responses to a 36 item questionnaire. SF-36 evaluated 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health from a range of 1 (better) to 5 (worst). The score for each section was an average of the individual question scores, which were scaled 0-100 (100=highest level of functioning). These 8 aspects were summarized as physical and mental component scores.
Time Frame: BL, Week (Wk) 24 and 48
Population: ITT-M2 population, n (number) = number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rituximab Escalated Dose Methotrexate: Participants received rituximab, 0.5 g, IV, on Days 1 and 15 and 1.0 g, IV, on Days 168 and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parenterally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose.
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 128 | 116 | 91
score on a scale
  Bodily Pain Score: BL (n=128,115,90) | 31.657 (7.5764) | 30.815 (6.5633) | 30.319 (6.2328)
  Bodily Pain Score: Wk 24 (n=118,108,87) | 39.709 (9.2218) | 38.875 (8.3432) | 42.736 (9.7885)
  Bodily Pain Score: Wk 48 (n=119,103,89) | 41.318 (9.2879) | 40.836 (8.6176) | 43.105 (9.4713)
  General Health Score: BL (n=127,116,90) | 34.850 (9.5814) | 34.692 (9.3289) | 34.025 (8.8533)
  General Health Score: Wk 24 (n=116,109,87) | 39.644 (9.8338) | 39.805 (10.2346) | 39.050 (10.4236)
  General Health Score: Wk 48 (n=118,101,89) | 41.138 (10.3191) | 41.555 (9.9892) | 40.427 (10.5756)
  Mental Health Score: BL (n=128,116,90) | 38.443 (12.4207) | 38.307 (11.9908) | 38.405 (11.1899)
  Mental Health Score: Wk 24 (n=118,108,87) | 43.506 (11.5661) | 43.209 (10.7315) | 43.955 (10.6107)
  Mental Health Score: Wk 48 (n=119,102,88) | 44.529 (11.7796) | 44.447 (11.9128) | 43.640 (11.5868)
  Physical Functioning Score: BL (n=127,116,91) | 28.826 (9.5523) | 28.223 (9.8730) | 29.896 (8.7899)
  Physical Functioning Score: Wk 24 (n=116,109,86) | 34.286 (11.1702) | 33.929 (11.3543) | 37.323 (10.5428)
  Physical Functioning Score: Wk 48 (n=118,103,89) | 35.291 (11.7203) | 35.318 (10.6680) | 38.547 (11.6649)
  Emotional Role Score: BL (n=127,115,90) | 33.719 (13.9238) | 32.217 (11.9819) | 32.167 (13.6914)
  Emotional Role Score: Wk 24 (n=117,109,87) | 39.665 (13.1752) | 37.406 (13.2790) | 39.928 (13.4008)
  Emotional Role Score: Wk 48 (n=118,102,88) | 40.429 (13.7266) | 39.644 (12.7514) | 39.800 (14.0611)
  Physical Role Score: BL (n=127,116,90) | 31.013 (9.5785) | 30.864 (8.7546) | 32.309 (9.4529)
  Physical Role Score: Wk 24 (n=117,109,86) | 37.694 (9.8439) | 36.977 (9.6325) | 39.027 (10.9050)
  Physical Role Score: Wk 48 (n=119,102,89) | 38.599 (10.9559) | 39.086 (9.6230) | 40.362 (10.1419)
  Social Functioning Score: BL (n=128,116,91) | 34.948 (11.6147) | 33.341 (11.3817) | 35.812 (12.2109)
  Social Functioning Score: Wk 24 (n=118,109,87) | 40.765 (10.5247) | 40.737 (10.4537) | 42.869 (10.8028)
  Social Functioning Score: Wk 48 (n=119,103,89) | 42.366 (11.1916) | 42.235 (11.0464) | 43.613 (11.3599)
  Vitality Score: BL (n=128,116,91) | 38.253 (10.2709) | 38.096 (9.5184) | 39.832 (10.2209)
  Vitality Score: Wk 24 (n=118,109,87) | 45.000 (10.7039) | 44.577 (11.1008) | 46.206 (10.0519)
  Vitality Score: Wk 48 (n=119,103,87) | 46.905 (10.5538) | 46.251 (10.8299) | 47.462 (11.3098)

8. Secondary Outcome: Change in SF-36 Score From BL
Description: as for outcome 7
Time Frame: BL, Weeks 24 and 48
Population: ITT-M2 population, n = number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 116 | 108 | 88
score on a scale
  Bodily Pain Score: Wk 24 (n=115,106,85) | 8.180 (9.7621) | 7.914 (8.7302) | 11.948 (10.2846)
  Bodily Pain Score: Wk 48 (n=116,101,87) | 9.815 (9.4616) | 9.323 (9.3335) | 12.712 (10.3962)
  General Health Score: Wk 24 (n=112,108,85) | 4.941 (8.8122) | 4.996 (8.7345) | 4.812 (8.1955)
  General Health Score: Wk 48 (n=115,100,87) | 6.470 (8.9736) | 6.340 (8.9124) | 6.241 (8.4496)
  Mental Health Score: Wk 24 (n=115,107,85) | 5.173 (10.5160) | 4.138 (11.5165) | 5.312 (8.1965)
  Mental Health Score: Wk 48 (n=116,101,86) | 6.607 (10.6356) | 4.979 (12.3225) | 4.939 (11.0695)
  Physical Functioning Score: Wk 24 (n=111,108,85) | 5.517 (7.6418) | 6.261 (8.2243) | 7.081 (9.4105)
  Physical Functioning Score: Wk 48 (n=114,102,88) | 6.529 (8.6382) | 6.318 (9.8785) | 8.577 (10.9439)
  Emotional Role Score: Wk 24 (n=113,108,85) | 5.951 (11.9256) | 4.571 (12.5182) | 7.180 (12.0934)
  Emotional Role Score: Wk 48 (n=114,101,86) | 6.445 (14.0187) | 6.350 (12.4357) | 7.142 (13.4771)
  Physical Role Score: Wk 24 (n=113,108,84) | 6.473 (9.1079) | 5.994 (9.7472) | 6.385 (9.6101)
  Physical Role Score: Wk 48 (n=115,101,87) | 7.347 (10.0663) | 7.493 (9.8317) | 7.873 (9.6133)
  Social Functioning Score: Wk 24 (n=115,108,86 | 5.786 (9.8861) | 7.070 (11.1663) | 6.722 (9.8518)
  Social Functioning Score: Wk 48 (n=116,102,88) | 7.382 (10.9376) | 7.807 (11.1880) | 7.713 (11.3046)
  Vitality Score: Wk 24 (n=115,108,86) | 6.796 (10.7057) | 6.495 (10.2488) | 6.534 (8.8644)
  Vitality Score: Wk 48 (n=116,102,86) | 9.088 (10.6821) | 7.479 (10.2350) | 7.200 (10.3652)

9. Secondary Outcome: Maximum Observed Serum Concentrations Following the 1st Infusion of Rituximab (Cfirst) in the 1st and 2nd Courses of Treatment in Micrograms Per mL (µg/mL)
Description: Cfirst values were estimated from rituximab serum concentrations by non-compartmental methods using the software WinNonlin Enterprise Version 5.2.
Time Frame: Days 1 and 15 (before infusion and 30 minutes following infusion) and Weeks 4, 8, 16, 24, 26, 28, 32, 40, and 48 or early withdrawal and at Weeks 24 and 48 of safety follow-up (1 year period following the completion of study treatment).
Population: ITT-M2 population, n = number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 121 | 112 | 91
µg/mL
  First Course (n=121,112,91) | 165 (42) | 163 (39) | 317 (94)
  Second Course (n=120,105,84) | 177 (41) | 345 (92) | 350 (86)

10. Secondary Outcome: Maximum Observed Serum Concentrations Following the 2nd Infusion of Rituximab (Csecond) in the 1st and 2nd Courses of Treatment in µg/mL
Description: Csecond values were estimated from rituximab serum concentrations by non-compartmental methods using the software WinNonlin Enterprise Version 5.2.
Time Frame: as for outcome 9
Population: ITT-M2 population, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 130 | 116 | 90
µg/mL
  First course (n=130,116,90) | 194 (65) | 190 (57) | 373 (116)
  Second course (n=121,107,88) | 209 (70) | 380 (139) | 392 (123)

11. Secondary Outcome: Terminal Elimination Half-Life (t1/2) in the 1st and 2nd Courses of Treatment in Days
Description: t1/2 values were estimated from rituximab serum concentrations by non-compartmental methods using the software WinNonlin Enterprise Version 5.2.
Time Frame: as for outcome 9
Population: ITT-M2 population, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 120 | 109 | 85
days
  First Course (n=120,109,85) | 16.04 (5.52) | 16.75 (6.64) | 17.67 (6.00)
  Second Course (n=116,99,85) | 19.62 (6.05) | 22.13 (6.48) | 21.42 (6.32)

12. Secondary Outcome: Peripheral Cluster of Differentiation (CD) 19 Positive (+) B Cell Count at BL in Cells Per Microliter (Cells/µL)
Description: Surface expression of CD19 was assessed by fluorescence-activated cell sorting (FACS) analysis as a marker of absolute B lymphocyte count.
Time Frame: BL
Population: ITT-M2 population. 7, 8, 3, 1, and 2 participants were not analyzed for this outcome measure from the Low Dose, Escalated Dose, High Dose, Placebo, and Decreased Dose groups, respectively.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 127 | 111 | 90 | 5 | 23
cells/µL | 183.6 (142.31) | 168.9 (94.98) | 205.3 (171.91) | 318.2 (174.62) | 235.4 (112.56)

13. Secondary Outcome: Percentage of Participants With Peripheral CD19+ B Cell Counts Above BL or the Lower Limit of Normal (LLN)
Description: Surface expression of CD19 was assessed by FACS analysis as a marker of absolute B lymphocyte count. The LLN was defined as < 80 cells/µL.
Time Frame: BL, Days 1 and 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: ITT-M2 population, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 127 | 114 | 91 | 6 | 24
percentage of participants
  Day 1 Postdose (n=118,109,85,5,23) | 0.8 | 0.0 | 2.4 | 0.0 | 8.7
  Day 15 Predose (n=127,114,87,5,24) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Day 15 Postdose (n=121,108,89,6,23) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Wk 4 (n=127,111,87,6,24) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Wk 8 (n=126,111,90,6,23) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Wk 16 (n=122,112,91,6,23) | 0.8 | 0.9 | 0.0 | 0.0 | 0.0
  Wk 24 (n=114,107,87,4,24) | 7.0 | 6.5 | 4.6 | 0.0 | 12.5
  Wk 28 (n=121,103,86,6,25) | 0.8 | 0.0 | 2.3 | 0.0 | 0.0
  Wk 32 (n=122,107,88,5,24) | 2.5 | 0.0 | 0.0 | 20.0 | 0.0
  Wk 40 (n=118,103,84,4,23) | 0.8 | 1.0 | 0.0 | 50.0 | 0.0
  Wk 48 (n=118,105,89,4,22) | 5.9 | 1.9 | 5.6 | 50.0 | 13.6

14. Secondary Outcome: Peripheral CD20+ B Cell Count in Cells/µL
Description: Surface expression of CD20 was assessed by FACS analysis as a marker of mature and memory B lymphocyte count.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: The safety analysis population (SAP) = ITT-M2 population, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 113 | 101 | 75
cells/µL
  BL Predose (n=113,97,75) | 184.8 (135.29) | 173.4 (99.18) | 218.1 (158.16)
  BL Postdose (n=105,94,71) | 0.2 (0.58) | 0.2 (0.49) | 0.2 (0.65)
  Day 15 Predose (n=112,101,75) | 0.6 (1.76) | 0.4 (0.74) | 0.3 (0.57)
  Day 15 Postdose (n=104,91,70) | 1.0 (7.35) | 0.2 (0.63) | 0.1 (0.39)
  Wk 4 (n=110,95,72) | 0.6 (3.21) | 0.2 (0.50) | 0.3 (0.74)
  Wk 8 (n=111,92,73) | 0.3 (0.64) | 4.9 (42.09) | 0.3 (0.86)
  Wk 16 (n=105,93,75) | 2.4 (8.02) | 3.0 (8.67) | 0.9 (3.15)
  Wk 24 (n=99,92,67) | 20.2 (53.56) | 15.2 (25.98) | 13.2 (23.96)
  Wk 28 (n=101,85,72) | 1.5 (12.14) | 1.1 (5.82) | 4.5 (20.59)
  Wk 32 (n=107,88,74) | 5.1 (33.42) | 1.1 (4.93) | 1.1 (6.88)
  Wk 40 (n=100,86,68) | 1.4 (5.44) | 1.7 (7.94) | 1.6 (9.11)
  Wk 48 (n=100,89,73) | 12.4 (26.89) | 4.4 (10.70) | 8.2 (22.12)

15. Secondary Outcome: Peripheral CD22+ B Cell Count in Cells/µL
Description: Surface expression of CD22 was assessed by FACS analysis as a marker of mature lymphocyte count.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 113 | 101 | 75
cells/µL
  BL Predose (n=113,97,75) | 188.0 (135.54) | 177.1 (98.69) | 221.6 (158.82)
  BL Postdose (n=105,94,71) | 24.5 (20.59) | 23.2 (17.39) | 29.0 (31.51)
  Day 15 Predose (n=112,101,75) | 5.0 (6.33) | 5.0 (6.03) | 5.1 (6.30)
  Day 15 Postdose (n=104,91,70) | 1.9 (1.92) | 1.9 (1.77) | 2.4 (3.23)
  Wk 4 (n=110,95,72) | 4.1 (5.61) | 3.8 (5.44) | 4.0 (7.73)
  Wk 8 (n=111,92,73) | 3.6 (5.14) | 8.4 (41.87) | 3.9 (6.03)
  Wk 16 (n=105,93,75) | 5.1 (8.60) | 6.1 (9.83) | 3.6 (5.94)
  Wk 24 (n=99,92,67) | 20.1 (32.29) | 17.6 (25.81) | 16.6 (25.70)
  Wk 28 (n=101,85,72) | 4.2 (13.16) | 4.0 (8.07) | 8.2 (21.96)
  Wk 32 (n=107,88,74) | 8.0 (33.71) | 3.7 (8.58) | 3.6 (8.51)
  Wk 40 (n=100,86,68) | 3.7 (6.92) | 3.5 (8.05) | 4.0 (10.01)
  Wk 48 (n=100,89,73) | 14.3 (26.88) | 6.3 (10.77) | 9.8 (22.24)

16. Secondary Outcome: Peripheral CD19+CD27+ B Cell Count in Cells/µL
Description: Simultaneous surface expression of CD19 and CD27 was assessed by FACS analysis as a marker of memory B lymphocyte count.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 113 | 99 | 75
cells/µL
  BL Predose (n=113,98,75) | 41.4 (41.79) | 42.2 (40.74) | 42.3 (33.71)
  BL Postdose (n=105,94,72) | 4.6 (2.85) | 5.1 (4.20) | 4.7 (3.40)
  Day 15 Predose (n=112,99,75) | 5.1 (4.65) | 4.5 (3.40) | 4.5 (2.83)
  Day 15 Postdose (n=103,89,70) | 3.0 (0.20) | 3.0 (0.24) | 3.0 (0.27)
  Wk 4 (n=110,92,74) | 4.6 (3.56) | 4.0 (2.70) | 4.6 (4.57)
  Wk 8 (n=110,92,75) | 4.6 (2.98) | 4.3 (2.51) | 4.6 (2.73)
  Wk 16 (n=104,93,75) | 5.5 (4.20) | 5.5 (4.39) | 4.9 (4.33)
  Wk 24 (n=97,91,67) | 6.8 (4.67) | 6.8 (5.95) | 7.1 (5.80)
  Wk 28 (n=101,86,72) | 5.3 (3.97) | 4.8 (3.54) | 4.1 (2.51)
  Wk 32 (n=105,88,73) | 5.7 (5.35) | 4.5 (3.38) | 5.3 (4.14)
  Wk 40 (n=99,84,67) | 5.6 (6.24) | 4.7 (3.41) | 4.9 (4.28)
  Wk 48 (n=96,87,70) | 5.4 (4.04) | 5.3 (4.11) | 6.5 (11.94)

17. Secondary Outcome: Peripheral CD19+CD27 Negative (-) B Cell Count in Cells/µL
Description: Surface expression of CD19 in the absence of CD27 expression was assessed by FACS analysis as a marker of naive B lymphocyte count.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 113 | 99 | 75
cells/µL
  BL Predose (n=113,98,75) | 141.1 (108.90) | 126.4 (75.00) | 179.3 (169.38)
  BL Postdose (n=105,94,72) | 16.7 (13.10) | 15.2 (9.5) | 19.3 (21.92)
  Day 15 Predose (n=112,99,75) | 10.2 (1.39) | 10.2 (0.94) | 10.2 (1.07)
  Day 15 Postdose (n=103,89,70) | 10.0 (0.00) | 10.0 (0.00) | 10.0 (0.00)
  Wk 4 (n=110,92,74) | 10.1 (0.90) | 10.1 (0.56) | 10.4 (1.68)
  Wk 8 (n=110,92,75) | 10.1 (0.49) | 10.1 (0.44) | 10.4 (1.77)
  Wk 16 (n=104,93,75) | 11.3 (6.65) | 11.7 (6.55) | 10.5 (2.04)
  Wk 24 (n=97,91,67) | 23.3 (25.11) | 21.7 (23.50) | 20.8 (20.89)
  Wk 28 (n=101,86,72) | 11.0 (9.15) | 10.5 (3.30) | 13.7 (19.34)
  Wk 32 (n=105,88,73) | 13.8 (27.58) | 10.9 (4.07) | 10.7 (5.86)
  Wk 40 (n=99,84,67) | 10.7 (4.33) | 11.3 (8.70) | 11.0 (7.59)
  Wk 48 (n=96,87,70) | 18.8 (22.13) | 13.0 (11.67) | 15.8 (18.69)

18. Secondary Outcome: Peripheral CD3+ T Cell Count in Cells/µL
Description: Surface expression of CD3 was assessed by FACS analysis as a marker of absolute T lymphocyte count. The normal range of CD3+ T cells was defined as 723-2737 cells/µL.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 127 | 114 | 91
cells/µL
  BL Predose (n=127,110,90) | 1262.1 (651.88) | 1229.6 (565.79) | 1319.7 (569.57)
  BL Postdose (n=118,109,85) | 237.8 (133.09) | 263.4 (167.58) | 226.9 (122.02)
  Day 15 Predose (n=127,114,87) | 1282.4 (587.75) | 1292.5 (589.57) | 1356.0 (604.98)
  Day 15 Postdose (n=121,108,89) | 302.5 (149.80) | 350.0 (220.23) | 343.3 (184.44)
  Wk 4 (n=127,111,87) | 1231.0 (585.60) | 1193.6 (505.68) | 1264.8 (508.87)
  Wk 8 (n=126,111,90) | 1262.8 (643.60) | 1317.3 (629.87) | 1296.0 (534.19)
  Wk 16 (n=122,112,91) | 1256.0 (580.95) | 1317.1 (605.57) | 1260.2 (562.16)
  Wk 24 (n=113,107,85) | 1332.1 (658.82) | 1297.1 (602.07) | 1314.9 (511.18)
  Wk 28 (n=120,101,86) | 1300.3 (670.68) | 1223.6 (505.72) | 1327.7 (590.38)
  Wk 32 (n=122,107,88) | 1318.8 (650.01) | 1286.0 (522.82) | 1312.6 (509.52)
  Wk 40 (n=118,103,84) | 1283.9 (620.88) | 1293.9 (559.38) | 1306.4 (508.49)
  Wk 48 (n=114,103,83) | 1280.6 (622.21) | 1251.8 (511.15) | 1315.8 (598.66)

19. Secondary Outcome: Change From BL in Peripheral CD3+ T Cell Count
Description: as for outcome 18
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 122 | 107 | 88
cells/µL
  BL Postdose (n=115,106,82) | -1000.6 (576.77) | -968.8 (539.80) | -1065.4 (513.18)
  Day 15 Predose (n=122,107,84) | 25.2 (478.94) | 40.8 (435.72) | 34.0 (463.99)
  Day 15 Postdose (n=116,102,86) | -952.6 (572.95) | -897.3 (535.33) | -965.9 (500.78)
  Wk 4 (n=122,105,84) | -31.9 (427.92) | -19.6 (450.67) | -53.3 (476.03)
  Wk 8 (n=121,105,87) | 3.4 (548.80) | 98.8 (496.83) | -23.6 (429.32)
  Wk 16 (n=117,105,88) | -24.5 (517.71) | 81.8 (436.08) | -47.4 (506.89)
  Wk 24 (n=109,100,82) | 78.1 (511.99) | 47.7 (448.72) | -0.8 (444.81)
  Wk 28 (n=115,94,84) | 41.4 (599.47) | 20.1 (379.99) | -0.4 (488.79)
  Wk 32 (n=116,99,85) | 47.9 (557.67) | 51.2 (412.36) | -18.4 (439.47)
  Wk 40 (n=113,96,81) | 33.5 (517.70) | 65.1 (511.46) | -12.7 (421.39)
  Wk 48 (n=110,96,80) | -9.4 (538.12) | 20.3 (431.58) | -12.4 (502.20)

20. Secondary Outcome: Peripheral CD4+ T Cell Count in Cells/µL
Description: Surface expression of CD4 was assessed by FACS analysis as a marker of T helper cell count. The normal range of CD4+ T cells was defined as 404-1612 cells/µL.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 127 | 114 | 91
cells/µL
  BL Predose (n=127,110,90) | 900.4 (500.42) | 876.7 (398.85) | 953.6 (462.18)
  BL Postdose (n=118,109,85) | 130.2 (81.65) | 145.9 (86.22) | 129.8 (75.17)
  Day 15 Predose (n=127,114,87) | 920.2 (468.01) | 930.1 (424.72) | 991.9 (504.25)
  Day 15 Postdose (n=121,108,89) | 165.4 (92.96) | 196.7 (124.38) | 196.9 (132.65)
  Wk 4 (n=127,111,87) | 880.5 (456.63) | 859.7 (373.69) | 917.9 (431.93)
  Wk 8 (n=126,111,90) | 903.3 (514.94) | 949.2 (462.71) | 950.5 (458.27)
  Wk 16 (n=122,112,91) | 889.2 (436.84) | 937.8 (450.52) | 910.1 (472.95)
  Wk 24 (n=113,107,85) | 969.6 (553.17) | 918.4 (434.08) | 948.2 (418.09)
  Wk 28 (n=120,101,86) | 936.6 (539.94) | 870.2 (373.17) | 967.0 (496.62)
  Wk 32 (n=122,107,88) | 939.0 (515.71) | 911.6 (404.40) | 950.9 (439.04)
  Wk 40 (n=118,103,84) | 908.7 (478.40) | 901.9 (383.73) | 942.6 (422.23)
  Wk 48 (n=114,103,83) | 908.2 (477.46) | 889.8 (378.08) | 952.7 (487.98)

21. Secondary Outcome: Change From BL in Peripheral CD4+ T Cell Count
Description: as for outcome 20
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 122 | 107 | 88
cells/µL
  BL Postdose (n=115,106,82) | -744.6 (454.55) | -738.1 (393.02) | -801.2 (416.45)
  Day 15 Predose (n=122,107,84) | 24.3 (355.22) | 38.9 (306.89) | 36.0 (359.92)
  Day 15 Postdose (n=116,102,86) | -732.2 (449.99) | -696.5 (392.37) | -749.4 (401.01)
  Wk 4 (n=122,105,84) | -16.1 (330.20) | -4.2 (345.57) | -36.2 (368.83)
  Wk 8 (n=121,105,87) | 7.9 (418.85) | 84.1 (370.64) | -4.4 (343.31)
  Wk 16 (n=117,105,88) | -24.3 (377.76) | 64.0 (349.16) | -33.4 (407.52)
  Wk 24 (n=109,100,82) | 72.6 (395.29) | 37.3 (312.15) | -0.7 (336.19)
  Wk 28 (n=115,94,84) | 42.8 (446.65) | 13.5 (276.55) | 7.4 (377.73)
  Wk 32 (n=116,99,85) | 38.4 (419.78) | 39.2 (305.18) | -8.4 (337.42)
  Wk 40 (n=113,96,81) | 14.9 (375.97) | 39.5 (356.89) | -6.4 (331.87)
  Wk 48 (n=110,96,80) | -8.5 (399.48) | 15.2 (320.98) | -10.1 (366.44)

22. Secondary Outcome: Peripheral CD8+ T Cell Count in Cells/µL
Description: Surface expression of CD8 was assessed by FACS analysis as a marker of cytotoxic T lymphocyte count. The normal range of CD8+ T cells was defined as 220-1129 cells/µL.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 127 | 114 | 91
cells/µL
  BL Predose (n=127,110,90) | 361.8 (231.86) | 352.6 (228.43) | 364.9 (181.22)
  BL Postdose (n=118,109,85) | 106.8 (70.64) | 118.6 (104.11) | 98.1 (70.68)
  Day 15 Predose (n=127,114,87) | 358.8 (196.37) | 360.9 (232.26) | 359.7 (174.12)
  Day 15 Postdose (n=121,108,89) | 134.0 (79.79) | 152.6 (130.11) | 145.6 (95.64)
  Wk 4 (n=127,111,87) | 348.4 (202.67) | 330.7 (197.94) | 341.9 (164.61)
  Wk 8 (n=126,111,90) | 357.3 (199.77) | 367.9 (239.39) | 342.3 (159.31)
  Wk 16 (n=122,112,91) | 365.1 (220.35) | 377.8 (227.32) | 344.2 (169.67)
  Wk 24 (n=113,107,85) | 359.1 (189.24) | 382.0 (241.73) | 363.3 (184.04)
  Wk 28 (n=120,101,86) | 359.9 (208.91) | 353.7 (221.13) | 357.3 (182.90)
  Wk 32 (n=122,107,88) | 372.3 (213.84) | 372.7 (211.86) | 359.9 (169.32)
  Wk 40 (n=118,103,84) | 367.8 (215.21) | 386.7 (260.49) | 356.7 (166.19)
  Wk 48 (n=114,103,83) | 365.9 (218.78) | 357.8 (210.51) | 355.5 (178.67)

23. Secondary Outcome: Change From BL in Peripheral CD8+ Cell Count
Description: as for outcome 22
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 122 | 107 | 88
cells/µL
  BL Postdose (n=115,106,82) | -256.2 (190.92) | -229.0 (183.97) | -262.3 (148.57)
  Day 15 Predose (n=122,107,84) | -1.5 (140.66) | 2.6 (167.12) | -5.0 (122.68)
  Day 15 Postdose (n=116,102,86) | -222.4 (180.50) | -201.4 (176.30) | -215.5 (140.77)
  Wk 4 (n=122,105,84) | -17.3 (127.14) | -18.0 (128.02) | -17.6 (124.74)
  Wk 8 (n=121,105,87) | -6.6 (157.14) | 16.3 (148.14) | -21.3 (101.94)
  Wk 16 (n=117,105,88) | -1.2 (176.58) | 18.0 (117.74) | -16.3 (114.90)
  Wk 24 (n=109,100,82) | 2.1 (150.31) | 14.3 (160.58) | 0.4 (130.37)
  Wk 28 (n=115,94,84) | -3.5 (183.31) | 7.2 (139.69) | -7.3 (130.24)
  Wk 32 (n=116,99,85) | 3.6 (163.20) | 11.6 (144.92) | -8.6 (129.83)
  Wk 40 (n=113,96,81) | 11.9 (174.03) | 22.3 (197.32) | -8.5 (112.07)
  Wk 48 (n=110,96,80) | -6.1 (168.67) | 2.2 (143.87) | -10.1 (150.14)

24. Secondary Outcome: Peripheral CD16+56+ Natural Killer (NK) Cell Count in Cells/µL
Description: Simultaneous surface expression of CD16 and CD56 was assessed by FACS analysis as a marker of NK cell count.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 127 | 114 | 91
cells/µL
  BL Predose (n=127,110,90) | 172.3 (102.58) | 173.5 (100.55) | 174.3 (99.82)
  BL Postdose (n=118,109,85) | 99.2 (51.46) | 111.7 (56.35) | 92.4 (52.96)
  Day 15 Predose (n=127,114,87) | 175.7 (95.76) | 180.6 (114.27) | 168.8 (84.38)
  Day 15 Postdose (n=121,108,89) | 170.8 (100.96) | 181.8 (103.36) | 173.7 (96.23)
  Wk 4 (n=127,111,87) | 180.1 (103.51) | 182.0 (110.95) | 173.2 (94.15)
  Wk 8 (n=126,111,90) | 197.7 (107.89) | 189.3 (105.93) | 177.8 (92.23)
  Wk 16 (n=122,112,91) | 201.7 (115.66) | 193.8 (120.85) | 184.1 (87.33)
  Wk 24 (n=113,107,85) | 188.8 (93.43) | 201.8 (120.24) | 182.6 (99.76)
  Wk 28 (n=120,101,86) | 203.4 (120.70) | 200.1 (119.07) | 200.8 (114.49)
  Wk 32 (n=122,107,88) | 212.5 (127.77) | 219.0 (130.92) | 193.8 (93.87)
  Wk 40 (n=118,103,84) | 222.4 (145.80) | 213.0 (127.08) | 214.8 (122.52)
  Wk 48 (n=114,103,83) | 208.4 (117.23) | 216.2 (128.45) | 212.2 (111.62)

25. Secondary Outcome: Change From BL in Peripheral CD16+56+ Cell Count
Description: Simultaneous surface expression of CD16 and CD56 was assessed by FACS analysis as a marker of NK cell count.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 122 | 107 | 88
cells/µL
  BL Postdose (n=115,106,82) | -72.2 (92.33) | -60.5 (93.63) | -83.2 (84.98)
  Day 15 Predose (n=122,107,84) | 4.0 (72.79) | 4.5 (74.48) | -1.4 (64.87)
  Day 15 Postdose (n=116,102,86) | -0.2 (91.95) | 8.8 (104.11) | -2.7 (84.49)
  Wk 4 (n=122,105,84) | 8.8 (81.85) | 15.6 (80.56) | 3.4 (79.93)
  Wk 8 (n=121,105,87) | 25.7 (88.56) | 15.1 (82.02) | 4.8 (61.94)
  Wk 16 (n=117,105,88) | 29.1 (96.16) | 17.2 (73.16) | 12.3 (80.04)
  Wk 24 (n=109,100,82) | 13.2 (89.73) | 28.8 (86.61) | 8.0 (76.78)
  Wk 28 (n=115,94,84) | 30.3 (103.95) | 29.5 (95.65) | 24.8 (81.95)
  Wk 32 (n=116,99,85) | 41.0 (109.60) | 39.8 (90.37) | 19.0 (82.51)
  Wk 40 (n=113,96,81) | 53.6 (125.06) | 38.8 (101.55) | 40.6 (90.44)
  Wk 48 (n=110,96,80) | 34.7 (94.33) | 39.8 (87.49) | 38.9 (85.59)

26. Secondary Outcome: Percentage of Participants With Total Immunoglobin (Ig), IgA, IgG, and IgM Results Below the LLN
Description: The LLNs for total Ig, IgA, IgG, and IgM were defined as 6.75 grams per liter (g/L), 0.70 g/L, 65 g/L, and 0.40 g/L, respectively.
Time Frame: BL, Weeks 24 and 48
Population: ITT-M2 population, n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 131 | 113 | 93 | 6 | 25
percentage of participants
  BL, total Ig <LLN (n=131,113,93,6,25) | 0.8 | 0.9 | 1.1 | 0.0 | 0.0
  BL, total IgA <LLN (n=131,113,93,6,25) | 0.8 | 0.9 | 2.2 | 0.0 | 0.0
  BL, total IgG <LLN (n=131,113,93,6,25) | 2.3 | 0.9 | 2.2 | 0.0 | 0.0
  BL, total IgM <LLN (n=131,113,93,6,25) | 0.8 | 0.0 | 1.1 | 0.0 | 4.0
  Wk 24, total Ig <LLN (n=117,109,83,4,24) | 0.9 | 0.9 | 0.0 | 0.0 | 0.0
  Wk 24, total IgA <LLN (n=117,109,83,4,24) | 0.0 | 0.9 | 1.2 | 0.0 | 0.0
  Wk 24, total IgG <LLN (n=117,109,83,4,24) | 0.9 | 0.9 | 0.0 | 0.0 | 0.0
  Wk 24, total IgM <LLN (n=117,109,83,4,24) | 7.7 | 7.3 | 6.0 | 0.0 | 16.7
  Wk 48, total Ig <LLN (n=117,105,89,4,22) | 0.9 | 0.0 | 0.0 | 0.0 | 4.5
  Wk 48, total IgA <LLN (n=117,105,89,4,22) | 1.7 | 1.0 | 2.2 | 0.0 | 0.0
  Wk 48, total IgG <LLN (n=117,105,89,4,22) | 1.7 | 0.0 | 0.0 | 0.0 | 4.5
  Wk 48, total IgM <LLN (n=117,105,89,4,22) | 13.7 | 13.3 | 10.1 | 0.0 | 18.2

27. Secondary Outcome: Percentage of Participants Who Were Rheumatoid Factor (RF) - Seronegative
Description: Percentage of participants who were RF seropositive at BL who became RF seronegative over the course of the study. RF seropositive status was defined as RF ≥ 20 international units (IU) per mL. RF seronegative status was defined as RF < 20 IU/mL.
Time Frame: BL, Weeks 8, 24, and 48
Population: RF seropositive participants from the ITT-M2 population, n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 93 | 84 | 60
percentage of participants
  Wk 8 (n=93,84,60) | 9.7 | 9.5 | 5.0
  Wk 24 (n=83,79,56) | 22.9 | 21.5 | 16.1
  Wk 48 (n=85,78,60) | 30.6 | 30.8 | 23.3

28. Secondary Outcome: Anti-Cyclic Citrullinated Peptide (CCP) Antibody Titers at BL in Units Per mL (U/mL)
Time Frame: BL
Population: SAP. 3, 3, and 2 participants were not analyzed for this outcome measure from the Low Dose, Escalated Dose, and High Dose, groups, respectively.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 131 | 116 | 91 | 6 | 25
U/mL | 205.39 (374.203) | 179.01 (255.251) | 263.61 (477.554) | 184.77 (304.169) | 310.94 (334.849)

29. Secondary Outcome: Change From BL in Anti-CCP Antibody Titers in U/mL
Time Frame: Weeks 8, 24, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 127 | 112 | 87 | 6 | 24
U/mL
  Wk 8 (n=127,112,85,6,24) | -42.97 (94.873) | -46.84 (140.589) | -70.39 (265.694) | -33.80 (58.443) | -18.67 (54.228)
  Wk 24 (n=117,107,82,4,24) | -68.23 (158.951) | -56.76 (144.256) | -72.96 (219.466) | -70.33 (149.881) | -64.32 (89.763)
  Wk 48 (n=116,102,87,4,22) | -72.99 (151.086) | -82.51 (223.577) | -127.21 (307.981) | -28.98 (42.881) | -81.57 (167.012)

30. Secondary Outcome: Percentage of Participants With Complement Component 3 (C3) Protein Level ≤ LLN
Description: The LLN for C3 protein was defined as <0.9 grams per liter (g/L).
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 127 | 115 | 88
percentage of participants
  BL Predose (n=127,108,86) | 3.1 | 0.9 | 1.2
  BL Postdose (n=122,109,87) | 3.3 | 2.8 | 5.7
  Day 15 Predose (n=124,115,84) | 2.4 | 0.9 | 2.4
  Day 15 Postdose (n=122,113,82) | 0.8 | 0.0 | 2.4
  Week 4 (n=121,113,83) | 3.3 | 0.0 | 1.2
  BL Pre Retreatment (n=121,105,88) | 6.6 | 1.9 | 3.4
  BL Post Retreatment (n=118,103,82) | 4.2 | 2.9 | 7.3
  Day 15 Pre Retreatment (n=120,105,86) | 6.7 | 1.9 | 7.0
  Day 15 Post Retreatment (n=119,107,88) | 5.9 | 4.7 | 8.0

31. Secondary Outcome: Change From BL in Complement C3 Protein Level in g/L
Description: The LLN of C3 protein was defined as <0.9 g/L.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 120 | 105 | 84
g/L
  BL Postdose (n=119,102,84) | -0.0469 (0.17761) | -0.0563 (0.16277) | -0.0802 (0.12774)
  Day 15 Predose (n=120,105,80) | -0.0423 (0.20915) | -0.0143 (0.17514) | -0.0773 (0.17876)
  Day 15 Postdose (n=118,104,79) | -0.0413 (0.18365) | -0.0235 (0.19255) | -0.1094 (0.21860)
  Wk 4 (n=118,105,78) | -0.0137 (0.22743) | 0.0279 (0.20724) | -0.0596 (0.18186)
  BL Pre Retreatment (n=115,98,83) | -0.0621 (0.21365) | -0.0225 (0.20578) | -0.0864 (0.19814)
  BL Post Retreatment (n=113,97,78) | -0.0889 (0.21974) | -0.0673 (0.21150) | -0.1395 (0.21823)
  Day 15 Pre Retreatment (n=115,97,81) | -0.0953 (0.20329) | -0.0580 (0.26221) | -0.1374 (0.19296)
  Day 15 Post Retreatment (n=113,99,82) | -0.1048 (0.20255) | -0.0979 (0.23505) | -0.1533 (0.21412)

32. Secondary Outcome: Change From BL in Activated Complement Component 3a (C3a) Protein Level in g/L
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 27 | 21 | 22
g/L
  BL Postdose (n=27,21,22) | -326.9 (3990.88) | -92.8 (836.55) | 1319.9 (5104.05)
  Day 15 Predose (n=18,10,14) | -1176.8 (4494.98) | -17.1 (389.94) | 1054.1 (5409.76)
  Day 15 Postdose (n=18,10,14) | -1117.7 (4347.64) | -285.4 (403.44) | -164.9 (740.91)
  Wk 4 (n=14,9,11) | 103.9 (749.79) | -124.2 (921.23) | -142.4 (504.95)

33. Secondary Outcome: Percentage of Participants With Complement Component 4 (C4) Protein Level ≤ LLN
Description: The LLN of C4 protein was defined as < 0.1 g/L.
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 127 | 115 | 88
percentage of participants
  BL Predose (n=127,108,86) | 2.4 | 0.0 | 1.2
  BL Postdose (n=122,109,87) | 4.9 | 0.9 | 2.3
  Day 15 Predose (n=124,115,83) | 2.4 | 0.0 | 2.4
  Day 15 Postdose (n=121,113,81) | 2.5 | 0.0 | 1.2
  Wk 4 (n=121,111,81) | 1.7 | 0.0 | 2.5
  BL Pre Retreatment (n=121,105,88) | 1.7 | 1.0 | 1.1
  BL Post Retreatment (n=118,103,81) | 1.7 | 1.0 | 1.2
  Day 15 Pre Retreatment (n=120,105,86) | 1.7 | 0.0 | 1.2
  Day 15 Post Retreatment (n=119,107,88) | 2.5 | 0.9 | 1.1

34. Secondary Outcome: Change From BL in Complement C4 Protein Level in g/L
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 120 | 105 | 84
g/L
  BL Postdose (n=119,102,84) | -0.0187 (0.04950) | -0.0170 (0.04048) | -0.0220 (0.02710)
  Day 15 Predose (n=120,105,80) | -0.0139 (0.06109) | -0.0089 (0.04479) | -0.0230 (0.04330)
  Day 15 Postdose (n=117,104,79) | -0.0126 (0.05330) | -0.0071 (0.04819) | -0.0320 (0.04947)
  Wk 4 (n=118,104,78) | 0.0020 (0.06441) | 0.0069 (0.05476) | -0.0020 (0.08212)
  BL Pre Retreatment (n=115,98,83) | 0.0046 (0.06671) | 0.0214 (0.06848) | 0.0128 (0.12884)
  BL Post Retreatment (n=113,97,77) | -0.0017 (0.05998) | 0.0064 (0.05432) | -0.0068 (0.05746)
  Day 15 Pre Retreatment (n=115,97,81) | -0.0049 (0.06120) | 0.0138 (0.12093) | -0.0142 (0.05015)
  Day 15 Post Retreatment (n=113,99,82) | -0.0079 (0.06431) | -0.0014 (0.05706) | -0.0168 (0.05079)

35. Secondary Outcome: Change From BL in Activated Complement Component 4a (C4a) Protein Level in g/L
Time Frame: BL, Day 15, Weeks 4, 8, 16, 24, 28, 32, 40, and 48
Population: SAP, n = number of participants assessed for the given parameter at the specified timepoint
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate
Number analyzed (Participants) | 26 | 21 | 22
g/L
  BL Postdose (n=26,21,22) | -1424.3 (3801.86) | -480.1 (3137.12) | -3749.1 (13498.79)
  Day 15 Predose (n=18,10,14) | -971.3 (3149.08) | 3004.9 (10300.68) | 3.5 (1832.62)
  Day 15 Postdose (n=18,10,14) | -1885.3 (2458.08) | -333.0 (706.11) | -1011.1 (1574.01)
  Wk 4 (n=14,8,10) | 629.8 (5993.96) | 260.4 (1450.40) | 109.8 (1566.68)

36. Secondary Outcome: Percentage of Participants With Positive Human Anti-Chimeric Antibody (HACA) Titers
Description: A participant was defined as being HACA positive if the HACA serum level was ≥ 5 relative units (RU) per mL and the physician comment read that participant was "immunodepletable with rituximab".
Time Frame: BL, Weeks 24 and 48
Population: SAP, n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 131 | 115 | 91 | 6 | 25
percentage of participants
  BL (n=131,115,91,6,25) | 0.0 | 0.9 | 0.0 | 0.0 | 0.0
  Wk 24 (n=118,109,86,4,24) | 5.1 | 7.3 | 2.3 | 0.0 | 0.0
  Wk 48 (n=115,104,87,4,22) | 4.3 | 1.0 | 2.3 | 25.0 | 0.0

37. Secondary Outcome: Percentage of Participants With a Change From BL by Category in Anti-Nuclear Antibodies (ANA) Titers
Description: ANA titers were obtained by the following serum dilution schema: negative = negative, borderline = 1 diluted to (:) 40 or 1:80, and positive ≥ 1:160. The change categories were defined for the change from BL to Weeks 24 and 48 according to this schema. Negative to borderline was defined as any change from negative to borderline as no dilution is given for negative results. Negative to positive was defined as at least a two-fold positive change in dilution from BL. Borderline to negative was defined as any change from borderline to negative as no dilution is given for negative results. Borderline to positive was defined as at least a two-fold positive change in dilution from BL. Positive to borderline was defined as at least a two-fold negative change in dilution from BL. Positive to negative was defined as at least a two-fold negative change in dilution from BL. Unchanged was defined as any difference in dilution less than two-fold.
Time Frame: BL, Weeks 24 and 48
Population: SAP, n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 113 | 107 | 86 | 4 | 24
percentage of participants
  Wk 24, Negative to Borderline (n=113,107,80,4,24) | 7.1 | 1.9 | 7.5 | 0.0 | 4.2
  Wk 24, Borderline to Negative (n=113,107,80,4,24) | 14.2 | 16.8 | 11.3 | 25.0 | 0.0
  Wk 24, Borderline to Positive (n=113,107,80,4,24) | 0.0 | 0.9 | 1.3 | 0.0 | 0.0
  Wk 24, Positive to Borderline (n=113,107,80,4,24) | 0.9 | 0.0 | 6.3 | 0.0 | 0.0
  Wk 24, Positive to Negative (n=113,107,80,4,24) | 0.0 | 0.9 | 1.3 | 0.0 | 0.0
  Wk 24, Unchanged (n=113,107,80,4,24) | 77.9 | 79.4 | 72.5 | 75.0 | 95.8
  Wk 48, Negative to Borderline (n=112,102,86,4,22) | 2.7 | 2.0 | 2.3 | 0.0 | 0.0
  Wk 48, Borderline to Negative (n=112,102,86,4,22) | 23.2 | 24.5 | 16.3 | 50.0 | 9.1
  Wk 48, Borderline to Positive (n=112,102,86,4,22) | 0.0 | 1.0 | 0.0 | 0.0 | 0.0
  Wk 48, Positive to Borderline (n=112,102,86,4,22) | 5.4 | 3.9 | 7.0 | 0.0 | 4.5
  Wk 48, Positive to Negative (n=112,102,86,4,22) | 4.5 | 2.0 | 3.5 | 0.0 | 0.0
  Wk 48, Unchanged (n=112,102,86,4,22) | 64.3 | 66.7 | 70.9 | 50.0 | 86.4

38. Secondary Outcome: Percentage of Participants With Positive Recall Antigen Antibody Titers
Description: A positive titer result to recall antigens was defined as a serum antibody level equal to or above the following protective levels: tetanus toxoid ≥ 0.1 IU/mL, influenza A > 12 U/mL, influenza B > 12 U/mL, and streptococcus (S.) pneumococcus ≥ 1.0 mg/L.
Time Frame: BL, Weeks 24 and 48
Population: SAP, n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Groups:
- Rituximab Low Dose + Methotrexate: Participants received rituximab, 0.5 g, IV, on Days 1, 15, 168, and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parentally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose.
- Rituximab Escalated Dose + Methotrexate: Participants received rituximab, 0.5 g, IV, on Days 1 and 15 and 1.0 g, IV, on Days 168 and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parentally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose.
- Rituximab High Dose + Methotrexate: Participants received rituximab, 1.0 g, IV, on Days 1, 15, 168, and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parentally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose.
- Rituximab/Placebo + Methotrexate: Participants received rituximab, 1.0 g, IV, on Days 1 and 15, and a placebo, IV, on Days 168 and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parentally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose. This treatment group was not part of the planned analysis and was not analyzed for all outcomes measures since they did not receive the planned treatment.
- Rituximab Decreased Dose + Methotrexate: Participants received rituximab, 1.0 g, IV, on Days 1 and 15 and 0.5 g, IV, on Days 168 and 182. Participants also received methylprednisolone 100 mg, IV, by slow infusion, which was completed at least 30 minutes prior to each infusion of rituximab Days 1, 15, 168, and 182. Participants also received methotrexate 10-25 mg/mL, PO or parentally, as prescribed by the treating physician and in accordance with the local label. Participants also received a stable dose of folate ≥ 5 mg/week given either as a single dose or as a divided weekly dose. This treatment group was not part of the planned analysis and was not analyzed for all outcomes measures since they did not receive the planned treatment.
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Number analyzed (Participants) | 131 | 115 | 91 | 6 | 25
percentage of participants
  Rubella, Day 1 Predose (n=125,110,88,6,25) | 94.4 | 98.2 | 89.8 | 100.0 | 92.0
  Rubella, Wk 24 (n=114,107,82,4,24) | 93.9 | 97.2 | 90.2 | 100.0 | 91.7
  Rubella, Wk 48 (n=112,100,88,4,21) | 94.6 | 97.0 | 89.8 | 100.0 | 95.2
  S. Pneumococcus, Day 1 Predose (n=130,114,91,6,25) | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  S. Pneumococcus, Wk 24 (n=118,108,83,4,24) | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  S. Pneumococcus, Wk 48 (n=116,105,89,4,22) | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Tetanus Toxoid, Day 1 Predose (n=131,115,91,6,25) | 77.1 | 70.4 | 75.8 | 66.7 | 84.0
  Tetanus Toxoid, Wk 24 (n=118,107,83,4,24) | 72.0 | 69.2 | 73.5 | 75.0 | 62.5
  Tetanus Toxoid, Wk 48 (n=118,105,89,4,22) | 71.2 | 66.7 | 73.0 | 75.0 | 54.5
  Varicella, Day 1 Predose (n=129,114,88,6,25) | 94.6 | 94.7 | 97.7 | 100.0 | 96.0
  Varicella, Wk 24 (n=114,105,79,4,23) | 94.7 | 94.3 | 96.2 | 100.0 | 95.7
  Varicella, Wk 48 (n=114,101,87,4,22) | 94.7 | 94.1 | 96.6 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from BL to Week 4 of Safety Follow-Up (SFU), after which only serious AEs (SAEs) were collected for the remainder of the SFU. SFU was done 4, 12, 24, 36 and 48 weeks after withdrawal.
Description: The safety analysis group included all randomized participants who received at least 1 infusion of study medication.
Arm/Group | Rituximab Low Dose + Methotrexate | Rituximab Escalated Dose + Methotrexate | Rituximab High Dose + Methotrexate | Rituximab/Placebo + Methotrexate | Rituximab Decreased Dose + Methotrexate
Serious Adverse Events (participants affected / at risk) | 15/134 | 21/119 | 16/93 | 1/6 | 3/25
Other Adverse Events (participants affected / at risk) | 120/134 | 103/119 | 88/93 | 6/6 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Low Dose + Methotrexate (N=134) | Rituximab Escalated Dose + Methotrexate (N=119) | Rituximab High Dose + Methotrexate (N=93) | Rituximab/Placebo + Methotrexate (N=6) | Rituximab Decreased Dose + Methotrexate (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ocular vascular disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (General disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Device failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Low Dose + Methotrexate (N=134) | Rituximab Escalated Dose + Methotrexate (N=119) | Rituximab High Dose + Methotrexate (N=93) | Rituximab/Placebo + Methotrexate (N=6) | Rituximab Decreased Dose + Methotrexate (N=25)
Upper respiratory tract infection (Infections and infestations) | 39 | 37 | 28 | 1 | 6
Nasopharyngitis (Infections and infestations) | 31 | 25 | 27 | 4 | 7
Urinary tract infection (Infections and infestations) | 26 | 20 | 17 | 0 | 2
Bronchitis (Infections and infestations) | 23 | 14 | 17 | 0 | 5
Sinusitis (Infections and infestations) | 13 | 16 | 17 | 1 | 1
Influenza (Infections and infestations) | 18 | 11 | 12 | 1 | 2
Gastroenteritis (Infections and infestations) | 11 | 14 | 13 | 2 | 3
Pharyngitis (Infections and infestations) | 8 | 7 | 8 | 1 | 4
Lower respiratory tract infection (Infections and infestations) | 8 | 6 | 3 | 3 | 1
Rhinitis (Infections and infestations) | 7 | 9 | 5 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 11 | 5 | 1 | 0
Cystitis (Infections and infestations) | 6 | 7 | 5 | 0 | 0
Respiratory tract infection (Infections and infestations) | 5 | 7 | 4 | 0 | 1
Localised infection (Infections and infestations) | 2 | 3 | 5 | 0 | 1
Paronychia (Infections and infestations) | 2 | 6 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 4 | 0 | 2
Tooth abscess (Infections and infestations) | 3 | 3 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 2 | 0 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 43 | 33 | 30 | 4 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 10 | 10 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 15 | 5 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 8 | 3 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 8 | 6 | 5 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 7 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 5 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 58 | 45 | 36 | 4 | 9
Fall (Injury, poisoning and procedural complications) | 15 | 11 | 10 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 7 | 4 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 6 | 2 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 10 | 10 | 1 | 2
Nausea (Gastrointestinal disorders) | 13 | 6 | 14 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 11 | 13 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 5 | 6 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 5 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 7 | 4 | 4 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 5 | 6 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 5 | 1 | 1
Gastritis (Gastrointestinal disorders) | 4 | 3 | 3 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 10 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 5 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3 | 0 | 0
Headache (Nervous system disorders) | 15 | 10 | 14 | 1 | 2
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 3 | 5 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 4 | 4 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 4 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 13 | 14 | 14 | 0 | 6
Insomnia (Psychiatric disorders) | 11 | 4 | 1 | 1 | 2
Depression (Psychiatric disorders) | 5 | 9 | 4 | 0 | 0
Oedema peripheral (General disorders) | 8 | 5 | 6 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 4 | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 1 | 5 | 3 | 0 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 2 | 3 | 1 | 1
Seasonal allergy (Immune system disorders) | 3 | 1 | 0 | 1 | 0
Allergic oedema (Immune system disorders) | 1 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 8 | 7 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.